CLINICAL TRIAL: NCT05173870
Title: Wearable Device Remote Monitoring to Prevent Frailty Progression in Elderly: a Pilot Study
Brief Title: Remote Monitoring to Prevent Frailty Progression in the Elderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Collaborators: University of Molise (Other)
Responsible Party: Principal Investigator, Licia Iacoviello, Head of the Department of Epidemiology and Prevention, Neuromed IRCCS
Other Study IDs: DEP_022021
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Frailty; Elderly; Wearable Device
Keywords: Frailty; Wearable device; Elderly; Health status monitoring
MeSH Terms: conditions — Frailty | interventions — Wearable Electronic Devices

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During the baseline and follow-up visits (at 6 months), venous blood samples will be obtained by venipuncture from participants. Samples for this study will be analyzed to measure the general biochemical clinical parameters ( blood cells, inflammation biomarkers, lipid profile etc) and then they will be stored in straws containing the sample code and barcode in liquid nitrogen in a dedicated biobank at IRCCS NEUROMED.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Wearable device — The wearable devices has a biosensor able to daily collect,in a remote way, many biometric measurements such as: blood pressure, blood oxygenation, heart and respiratory rate

SUMMARY:
Frailty is a frequent condition in elderly, characterized by reduced physiologic reserve, leading to an increased risk for adverse events, such as disability, hospitalization, and death. In particular, it is a multidimensional disfunctional condition, including decreases in physiologic capacity in neurologic control (indicated by diminished ability to perform complex tasks), mechanical performance (e.g. diminished strength), and energy metabolism (e.g. decreased aerobic status due to cardiac or pulmonary diseases or both). All these factors lead to the worsening of quality of life. Focusing on the great impact of this condition in global population and the rising of social/health costs, related to this condition, frailty is earning a great interest from both at political level and European Community. For this reason, developing interventions programs aiming to prevent the progression of frailty towards the independence loss, it is considered a key objective for the improvement of the quality of life. In this context, this pilot study looks at the standardization of a study protocol to develop a useful model for enhancing local care in small population isolates, by remotely monitoring the health status of pre-frail subjects and improving the progression of the frailty condition, in order to support a healthy ageing for future investigation including a larger number of individuals.

DETAILED DESCRIPTION:
Frailty is a condition of increased vulnerability to stressors due to age-related declines in physiologic reserves across neuromuscular, metabolic, and immune systems. It is considered a medical geriatric syndrome with multiple causes and contributors and it is characterized by diminished strength, power and endurance. In general, therefore, frailty is considered to be a multifactorial dysfunctional framework which includes the physical, psychological, cognitive, economic and social spheres and which leads to a serious deterioration in the quality of life. Due to the great impact of this condition on quality of life, developing interventions programs aiming to prevent the progression of frailty towards the independence loss, it is considered a key objective to support an healthy ageing.

In this context, the primary aim of the present pilot study is to standardize a study protocol to develop a useful model to enhance local care in small population isolates, by remotely monitoring the health status of pre-frail subjects and to improve the progression of the frailty condition, in order to support a healthy ageing for future investigation including a larger number of individuals.

Additional aims:

* To quantify the timeframes necessary for the subjects recruiting and examination activities,including questionnaires and functional tests administration;
* To quantify the training time needed to explain the use of the wearable device to the recruited elderly individuals;
* To assess the responsiveness of pre-frail subjects, during the preliminary screening, the examination visit and the monitoring period (follow-up 6 months);
* To evaluate the compliance of pre-frail individuals with the use of the wearable device.

All men and women aged >= 65 years, resident a small mountain village (Salcito) in Molise region, Italy, will be invited to participate at the first examination, in order to evaluate their frailty condition, in a specific way their pre-frail/frail condition.

In the screening phase, in particular, it will be used the AGILE score to select the subjects to be included in the study. The questionnaire is a frailty tool that allows to quickly identify elderly, but also to investigate "multidimensional" frailty. It is built by selecting among the 40 items of the italian frailty index, the 10 ones most predictive of mortality. Therefore the questionnaire is composed by 10 items with a dychotomous answer (yes/no), in order to homogenously represent the four domains of frailty: physical, mental, nutrirional and socio-economic. After the preliminary screening, 30 elderly with pre-frailty will be randomly selected to be equipped with the wearable devices (such as smartband and smart-clothes ).The wearable devices have a biosensor able to daily collect,in a remote way, many biometric measurements such as: blood pressure, body temperature, heart and respiratory rate, posture and sleep quality.

During the baseline visit, the 30 pre-frail elderly will be trained to the use of the wearable devices. In addition, others questionnaires will be administered to collect information on their dietary habits, lifestyles, cognitive assessment and clinical history of the major chronic disease (CVD, cancer…). Additionally, during the baseline visit of recruited 30 pre-frail subjects, a venous blood sample will be collected. This will be used to measure biochemical and molecular parameters. In particular, samples will be analyzed to study potential biomarkers of pre-frailty/frailty condition. An aliquot of the biological sample will be stored in liquid nitrogen in a dedicated biobank of IRCCS (Istituto di Ricovero e Cura a Carattere Scientifico) NEUROMED, for any future molecular analysis.

Thanks to the wearable devices, individuals will be monitored constantly for six months, from a health point of view.

In the early stages of recruitment it will be possible to identify any critical issues in the training procedures of individuals over 65 recruited to use the wearable device.

During the six months period of monitoring, it will be possible to evaluate the compliance of subjects recruited to the wearable device use. In particular, it could be possible to evaluate the reliability of collected data thanks to the device and eventually make changes in operative procedures, when needed. If, during the monitoring, an abnormal parameter value will be observed, it will be communicated both to the subject and to his physician, with the aim of promoting a greater attention to personal health. In this way it could be possible to ensure a better quality of life. During six months, participants will be called back every other month, in order to evaluate the status of devices. After six months, participants will be called back for a follow-up visit, during which all the test, the questionnaires and the blood sample collection will be repeated to evaluate the potential impact of monitoring, on their condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Pre-Frail;
* Salcito (a small mountain village in Molise region) residents.

Exclusion Criteria:

* Age< 65 years;
* Individuals affected by physical or mental diseases, pacemaker or other medical device keeper who make the use of "wearable device" not possible or unable to complete functional tests.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: All men and women aged >= 65 years, resident in Salcito, a small mountain village in Molise region, Italy, will be invited to participate at the first examination, in order to evaluate their frailty condition, in a specific way their pre-frail/frail condition.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Study protocol assessment | From February 2022 to August 2023
  To standardize a study protocol to develop a useful model for enhancing local care in small population isolates, by remotely monitoring the health status of pre-frail subjects and improving the progression of the frailty condition in order to support a healthy ageing for future investigation including a larger number of individuals.

SECONDARY OUTCOMES:
Recruitment phase | From February 2022 to May 2022
  This pilot study will be performed to quantify the timeframes necessary for the recruitment of the elderly subjects and for the examination activities, including questionnaires and functional tests administration.
Training Phase | From February 2022 to May 2022
  This pilot study will be performed to quantify the training time needed to explain the use the wearable device to the recruited elderly individuals.
Pre-frail subjects responsiveness | From February 2022 to August 2022
  This pilot study want to assess the responsiveness (i.e.the active participation to the project) of pre-frail subjects.
  This aspect will be evaluated as follows:
  1. Affirmative response to the invitation to the screeening visit;
  2. Active participation and complete all the questionnaires during the examination visit;
  3. Collaboration and interactions with the researchers during the monitoring period (follow-up 6 months).
Wearable device compliance | From February 2022 to August 2022
  This pilot study want to evaluate the compliance of pre-frail individuals with the use of the wearable device.
  This aspect will be evaluated by monitoring the time during which subjects wear the device.
  If it is weared less than 5 days (20/24h) per week, it will be considered as a low compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Licia Iacoviello, MD, PhD, Principal Investigator — IRCCS Neuromed
Locations (2):
- Italy (2):
  - IRCCS INM Neuromed, Department of Epidemiology and Prevention, Pozzilli, IS
  - IRCCS Neuromed, Pozzilli, IS